CLINICAL TRIAL: NCT05427175
Title: Evaluation of the Effect of Narrowband Ultraviolet B Versus Methotrexate on Serum Chitotriosidase Level in Psoriasis.
Brief Title: Evaluation of the Effect of Narrowband UVB Versus Methotrexate on Serum Chitotriosidase Level in Psoriasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Shimaa Ali Hussien Ali, Principal investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 593/1/22
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Narrowband ultraviolet B (Active Comparator): Patients will receive 8 sessions of NB-UVB per month for 3 successive months
  Interventions: Radiation: Narrowband ultraviolet B
- Methotrexate (Active Comparator): Patients will receive 25 mg/1ml of methotrexate vial per week for 3 successive months
  Interventions: Drug: Methotrexate
- healthy individuals as control group (No Intervention)

INTERVENTIONS:
Radiation: Narrowband ultraviolet B — Patients will receive 8 sessions of NB-UVB per month for 3 successive months
  Other Names: NB-UVB
  Arms: Narrowband ultraviolet B
Drug: Methotrexate — Patients will receive 25 mg/1ml of methotrexate vial per week for 3 successive months
  Other Names: MTX
  Arms: Methotrexate

SUMMARY:
The aim of the study is to evaluate the effect of NB-UVB versus MTX on serum Chitotriosidase level in psoriatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe plaque psoriasis of any age and gender.

Exclusion Criteria:

* History of psoriasis treatment with systemic and biological agents prior to the study for at least 3 months.
* Pregnancy and lactation.
* Infections.
* Patients with chronic diseases: hepatic disorders, hematologic diseases, chronic renal failure or cancer.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Serum Chitotriosidase in psoriasis | 3 months
  Measurement of serum Chitotriosidase in psoriatic patients before and after treatment with NB-UVB versus MTX in comparison with healthy individuals, using ELISA (enzyme-linked immunosorbent assay).

SECONDARY OUTCOMES:
Treatment of psoriasis | 3 months
  Clinical evaluation: Assessment of disease severity will be performed by using psoriasis area severity index (PASI score) before and after treatment with NB-UVB in comparison with MTX.

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa A El Taieb, Study Chair — Faculty of medicine aswan university
Locations (1):
- Aswan University - Faculty of Medicine, Aswān, Aswan Governorate, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No